CLINICAL TRIAL: NCT00081289
Title: Randomized Phase II Trial Of Neoadjuvant Combined Modality Therapy For Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Chemoradiotherapy and Adjuvant Chemotherapy in Treating Patients Who Are Undergoing Surgical Resection for Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0247; CDR0000350136
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
Keywords: stage III rectal cancer; adenocarcinoma of the rectum; stage II rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Radiotherapy; Capecitabine; Irinotecan; Oxaliplatin; Surgical Procedures, Operative; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoadjuvant chemoradiation with irinotecan (Experimental): Patients receive neoadjuvant therapy comprising 45 Gy (1.8 Gy/fx) + 5.4 Gy boost (1.8 Gy/fx) radiation therapy (RT), oral capecitabine 1200mg/m^2/day 5 days/week during RT, and irinotecan 50 mg/m^2 IV for 1 hour days 1, 8, 22, 29. Surgery 4-8 weeks after RT. Postoperative chemotherapy beginning Day 1 postoperatively for nine 14-day cycles(folinic acid 400 mg/m^2 over 2 hours Day 1; 5-fluorouracil bolus 400 mg/m^2 IV push Day 1 plus 2400 mg/m^2 IV continuous infusion over 46 hours, beginning Day 1; and oxaliplatin 85 mg/m^2 IV over 2 hours Day 1) .
  Interventions: Radiation: Radiation Therapy; Drug: Capecitabine 1200 mg/m^2/day; Drug: Irinotecan; Procedure: Surgery; Drug: Folinic Acid; Drug: Fluorouracil; Drug: Oxaliplatin
- Neoadjuvant chemoradiation with oxaliplatin (Experimental): Patients receive neoadjuvant therapy comprising 45 Gy (1.8 Gy/fx) + 5.4 Gy boost (1.8 Gy/fx) radiation therapy (RT), oral capecitabine 1650mg/m^2/day 5 days/week during RT, and oxaliplatin 50 mg/m^2 IV for 2 hours days 1, 8, 15, 22, 29. Surgery 4-8 weeks after RT. Postoperative chemotherapy beginning Day 1 postoperatively for nine 14-day cycles(folinic acid 400 mg/m^2 over 2 hours Day 1; 5-fluorouracil bolus 400 mg/m^2 IV push Day 1 plus 2400 mg/m^2 IV continuous infusion over 46 hours, beginning Day 1; and oxaliplatin 85 mg/m^2 IV over 2 hours Day 1) .
  Interventions: Radiation: Radiation Therapy; Drug: Capecitabine 1650 mg/m^2/day; Drug: Oxaliplatin; Procedure: Surgery; Drug: Folinic Acid; Drug: Fluorouracil

INTERVENTIONS:
Radiation: Radiation Therapy — Pelvic radiation therapy given once daily 5 days a week for 6 weeks, 45 Gy in 25 fractions + boost of 5.4 Gy in 3 fractions for a total dose of 50.4 Gy.
Drug: Capecitabine 1650 mg/m^2/day — 825 mg/m^2 q12 hours (1650 mg/m^2/day) orally 5 days per week during radiotherapy.
  Arms: Neoadjuvant chemoradiation with oxaliplatin
Drug: Capecitabine 1200 mg/m^2/day — 600 mg/m^2 q12 hours(1200 mg/m^2/day) orally 5 days per week during radiotherapy.
  Arms: Neoadjuvant chemoradiation with irinotecan
Drug: Irinotecan — 50mg/m^2 IV over 1 hour on days 1, 8, 22, and 29
  Other Names: Irinotecan Hydrochloride
  Arms: Neoadjuvant chemoradiation with irinotecan
Drug: Oxaliplatin — 50mg/m^2 IV over 2 hours on days 1, 8, 15, 22, and 29
  Arms: Neoadjuvant chemoradiation with oxaliplatin
Procedure: Surgery — All patients will undergo surgery four to eight weeks following the completion of radiation therapy. The choice of procedure abdominoperineal resection (APR), low anterior resection (LAR), or LAR/coloanal anastomosis is at the discretion of the surgeon.
Drug: Folinic Acid — 400 mg/m^2 IV over 2 hours Day 1 (postoperatively) ,every 14 days, for nine 14-day cycles.
  Other Names: Leucovorin
Drug: Fluorouracil — 5-fluorouracil bolus 400 mg/m^2 IV push Day 1 (postoperatively), every 14 days, for nine 14-day cycles.
  5-fluorouracil infusion 2400 mg/m^2 IV continuous infusion over 46 hours, beginning day 1, every 14 days, for nine 14-day cycles.
  Other Names: 5-FU
Drug: Oxaliplatin — 85 mg/m^2 IV over 2 hours Day 1 (postoperatively), every 14 days, for nine 14-day cycles.

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Chemoradiotherapy (combining chemotherapy with radiation therapy) before surgery may shrink the tumor so that it can be removed. Giving chemotherapy after surgery may kill any remaining tumor cells.

PURPOSE: This randomized phase II trial is studying two different regimens of neoadjuvant chemoradiotherapy and adjuvant chemotherapy and comparing how well they work in treating patients who are undergoing surgical resection for locally advanced rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the pathologic complete response rate in patients with locally advanced rectal cancer undergoing surgical resection treated with 2 different regimens of neoadjuvant chemoradiotherapy and adjuvant chemotherapy.
* Evaluate the time to treatment failure and patterns of failure in patients treated with these regimens.
* Evaluate the incidence of hematologic and non-hematologic grade 3-4 toxicity (preoperatively, postoperatively, and overall) in patients treated with these regimens.
* Evaluate the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to clinical stage of tumor (T3 vs T4). Patients are randomized to 1 of 2 treatment arms.

Quality of life is assessed at baseline, within 1 week after completion of radiotherapy, within 1 week after completion of adjuvant chemotherapy (12 months), and then at 24 months.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the rectum originating at or below 12 cm from the anal verge without evidence of distant metastases
2. Patient must be 18 years of age or greater.
3. Potentially resectable en bloc based upon surgeon evaluation
4. Clinical stages T3 or T4, based upon endorectal ultrasound, or physical examination (only acceptable for T4 lesions).
5. Absolute neutrophil count of > 1500 per microliter and platelet count > 100,000 per microliter; aspartate aminotransferase (AST) and alkaline phosphatase < 2.5 X upper limit of normal (ULN), bilirubin < = 1.5 ULN, calculated creatinine clearance > 50 ml/min using Cockcroft-Gault formula:

   * CrCl male = (140 - age) x (wt. in kg) / (Serum Cr) x 72
   * CrCl female = 0.85 x (CrCl male)
6. Zubrod performance status 0-2
7. No history of other malignancies within 5 years, except non-melanoma skin cancer, in situ carcinoma of the cervix, or ductal carcinoma in situ of the breast. Previous invasive cancer permitted if disease free at least 5 years.
8. Signed study-specific informed consent prior to randomization

Exclusion Criteria:

1. Any evidence of distant metastasis
2. Synchronous primary colon carcinomas, except T1 lesions (full colonoscopy not required for enrollment)
3. Extension of malignant disease to the anal canal
4. Prior radiation therapy to the pelvis
5. Prior chemotherapy for malignancies
6. Pregnancy or lactation, (exclusion due to potential adverse effects of therapy). Women of childbearing potential with either a positive or no pregnancy test (serum or urine) at baseline. Women/men of childbearing potential not using a reliable and appropriate contraceptive method. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered to be of non-childbearing potential.) Patients will agree to continue contraception for 30 days from the date of the last study drug administration.
7. Serious, uncontrolled, concurrent infection(s).
8. Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
9. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
10. Evidence of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
11. Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
12. Major surgery within 4 weeks of the study treatment.
13. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
14. Known, existing uncontrolled coagulopathy.
15. No concurrent cimetidine allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2004-03; Primary Completion 2011-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal J. Meropol, MD, Principal Investigator — Fox Chase Cancer Center
Locations (5):
- United States (5):
  - University of California Davis Cancer Center, Sacramento, California
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania

REFERENCES:
- [Result] Wong SJ, Winter K, Meropol NJ, Anne PR, Kachnic L, Rashid A, Watson JC, Mitchell E, Pollock J, Lee RJ, Haddock M, Erickson BA, Willett CG. Radiation Therapy Oncology Group 0247: a randomized Phase II study of neoadjuvant capecitabine and irinotecan or capecitabine and oxaliplatin with concurrent radiotherapy for patients with locally advanced rectal cancer. Int J Radiat Oncol Biol Phys. 2012 Mar 15;82(4):1367-75. doi: 10.1016/j.ijrobp.2011.05.027. Epub 2011 Jul 19. PMID 21775070
- [Result] Wong SJ, Moughan J, Meropol NJ, et al.: Efficacy endpoints of RTOG 0247: A randomized phase II study of neoadjuvant capecitabine (C) and irinotecan (I) or C and oxaliplatin (O) with concurrent radiation therapy (RT) for locally advanced rectal cancer. [Abstract] J Clin Oncol 29 (Suppl 15): A-3517, 2011.

RESULTS

PARTICIPANT FLOW:
Groups:
- Neoadjuvant Chemoradiation With Irinotecan: Patients receive neoadjuvant therapy comprising radiotherapy (RT), 1200mg/m2/day oral capecitabine and irinotecan. Surgery 4-8 weeks after RT. Postoperative chemotherapy (folinic acid, fluorouracil, and oxaliplatin) 4-6 weeks after surgery.
- Neoadjuvant Chemoradiation With Oxaliplatin: Patients receive neoadjuvant therapy comprising radiotherapy, 1650mg/m2/day oral capecitabine and oxaliplatin. Surgery 4-8 weeks after RT. Postoperative chemotherapy (folinic acid, fluorouracil, and oxaliplatin) 4-6 weeks after surgery.
Period: Overall Study
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Started | 73 | 73
Primary Endpoint Population (First 48 eligible patients accrued per arm after the protocol amendment) | 48 | 48
General Analysis Population (Eligible participants enrolled after the protocol ammendment) | 52 | 52
Full AE Population (All eligible patients including those enrolled prior to protocol amendment) | 70 | 68
Surgery (Eligible patients enrolled after the protocol amendment who had surgery) | 47 | 51
Global Health Status Score at End of CR (EORTC QLQ-C30 Global Health Status (GHS) Score at baseline and end of chemoradiation (CR)) | 34 (European Organization for Research & Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ]) | 32
GHS at End of Post-op CT (EORTC QLQ-C30 GHS Score at baseline and end of post-operative chemotherapy (CT)) | 20 | 28
GHS at Two Years (EORTC QLQ-C30 GHS Score at baseline and two years) | 21 | 20
GI Symptom Score at End of CR (EORTC QLQ-CR38 Gastro-Intestinal (GI) Symptom Score at baseline and end of chemoradiation) | 34 | 33
GI Symptom Score at End of Post-op CT (EORTC QLQ-CR38 GI Symptom Score at baseline and end of post-operative chemotherapy) | 22 | 27
GI Symptom Score at Two Years (EORTC QLQ-CR38 GI Symptom Score at baseline and two years) | 21 | 20
Defecation Symptom Score at End of CR (EORTC QLQ-CR38 Defecation Symptom Score at baseline and end of chemoradiation) | 32 | 32
DS Score at End of Post-op CT (EORTC QLQ-CR38 Defecation Symptom (DS) Score at baseline and end of post-operative chemotherapy) | 12 | 14
Defecation Symptom Score at Two Years (EORTC QLQ-CR38 Defecation Symptom Score at baseline and two years) | 13 | 15
Completed (Subjects contributing any data to analysis are considered to have completed the study) | 52 | 52
Not Completed | 21 | 21
Not completed — Accrued prior to chemotherapy amendment | 18 | 17
Not completed — Ineligible / no protocol treatment | 3 | 4

BASELINE CHARACTERISTICS:
Population: Eligible patients enrolled after the protocol ammendment.
Groups:
- Neoadjuvant Chemoradiation With Irinotecan: Patients receive neoadjuvant therapy comprising radiotherapy, 1200mg/m2/day oral capecitabine and irinotecan. Surgery 4-8 weeks after RT. Postoperative chemotherapy (folinic acid, fluorouracil, and oxaliplatin) 4-6 weeks after surgery.
- Total: Total of all reporting groups
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Median (Full Range); unit: years] | 57 [27 to 78] | 56 [30 to 76] | 57 [27 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 33 | 38 | 71

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: A pathologic complete response (pCR) was defined as no evidence of residual cancer histologically; disease progression or death before surgery was considered less than pCR (even without surgical specimen). All cases were reviewed by the study's surgical oncology co-chair for the determination of pCR.
  Each arm was first analyzed alone. If the arm had 9 or more pCRs in 48 evaluable pts, then the null hypothesis (H0) of 10% pCR rate would be rejected in favor of the alternative hypothesis of 25%, providing 90% power with a two-sided 10% type I error rate. If both arms reject H0, then statistical selection theory would be used to choose the arm for further study in a phase III trial. If only one arm has acceptable pCR rate, then that arm would be pursued in a phase III trial.
Time Frame: After protocol surgery, approximately 10-16 weeks from randomization based on surgery occurring 4-8 weeks after chemoradiation
Population: For each arm the first 48 eligible enrolled after the protocol amendment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 48 | 48
percentage of participants | 10.4 [3.5 to 22.7] | 20.8 [10.5 to 35.0]

2. Secondary Outcome: Survival Rate at 4 Years
Description: Survival time is defined as time from registration/randomization to the date of death from any cause or last known follow-up (censored). Survival rates are estimated by the Kaplan-Meier method.
Time Frame: From randomization to four years
Population: Eligible patients enrolled after the protocol amendment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 52 | 52
percentage of participants | 85 [66 to 94] | 75 [60 to 85]

3. Secondary Outcome: Local-regional Failure Rate at 4 Years
Description: Local-regional failure is defined as any of the following: no clinical complete response (cCR) in the primary site and/or nodes at any time after treatment completion (persistence), recurrence and/or progression in the primary site and/or nodes after cCR, and nonprotocol surgery to the primary site after cCR. Time to local-regional failure is defined as time from randomization to date of failure, last known follow-up (censored), or death without local-regional failure (competing risk). Local-regional failure rates are estimated by the cumulative incidence method.
Time Frame: From randomization to four years
Population: Eligible patients enrolled after the protocol amendment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 52 | 52
percentage of participants | 16 [6 to 27] | 18 [7 to 28]

4. Secondary Outcome: Distant Failure Rate at 4 Years
Description: Time to distant failure is defined as time from randomization to date of the appearance of distant metastases, last known follow-up (censored), or death without distant failure (competing risk). Distant failure rates are estimated by the cumulative incidence method.
Time Frame: From randomization to four years
Population: Eligible patients enrolled after the protocol amendment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 52 | 52
percentage of participants | 24 [11 to 38] | 30 [17 to 43]

5. Secondary Outcome: Second Primary Rate at 4 Years
Description: Time to second primary is defined as time from randomization to date of the appearance of a second primary cancer, last known follow-up (censored), or death without second primary (competing risk). Second primary rates are estimated by the cumulative incidence method.
Time Frame: From randomization to four years
Population: Eligible patients enrolled after the protocol amendment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 52 | 52
percentage of participants | 2 [0 to 6] | 6 [0 to 13]

6. Secondary Outcome: Disease-free Survival Rate at 4 Years
Description: Disease-free survival time is defined as time from randomization to date of local-regional failure, the appearance of distant metastases, the appearance of a second primary failure, or date of death from any cause/ Disease-free survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive without failure are censored at the date of last contact.
Time Frame: From randomization to four years
Population: Eligible patients enrolled after the protocol amendment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 52 | 52
percentage of participants | 68 [52 to 80] | 62 [47 to 74]

7. Secondary Outcome: Number of Participants With Grade 3+ Treatment-related Adverse Events
Description: Highest grade adverse event per subject were counted. Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From start of treatment to end of follow-up. Maximum follow-up is 5.2 years.
Population: Eligible patients enrolled after the protocol amendment
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 52 | 52
Participants
  Hematologic | 20 | 19
  Non-Hematologic | 32 | 29
  Overall | 38 | 36

8. Secondary Outcome: Number of Participants With Grade 3+ Treatment-related Adverse Events Preoperatively
Description: as for outcome 7
Time Frame: From start of treatment to surgery, approximately 10-16 weeks from randomization based on surgery occurring 4-8 weeks after chemoradiation. If no surgery, then <= 90 days from start of treatment.
Population: Eligible patients enrolled after the protocol amendment
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 52 | 52
Participants
  Hematologic | 5 | 2
  Non-Hematologic | 11 | 14
  Overall | 14 | 14

9. Secondary Outcome: Number of Participants With Grade 3+ Treatment-related Adverse Events Postoperatively
Description: as for outcome 7
Time Frame: From post-surgery to before chemotherapy (CT), or within 60 days of surgery if no postoperative CT. Approximately 10-16 weeks to 14-22 weeks from randomization based on CT starting 4-6 weeks after surgery.
Population: Eligible patients enrolled after the protocol amendment who had surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 47 | 51
Participants
  Hematologic | 1 | 3
  Non-Hematologic | 9 | 9
  Overall | 9 | 10

10. Secondary Outcome: Tumor Marker Evaluation Using Preoperative Tissue Biopsy Specimens and Surgically Resected Tissue Specimens
Time Frame: End of study
Population: The data required for this analysis was not obtained and will not be obtained.
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in QLQ-C30 Global Health Status Score at Completion of Chemoradiation
Description: Global Health Status is calculated from two questions on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ]-C30. The question responses range from 1 "very poor" to 7 "excellent" such that a higher response indicates better quality of life (QOL). The mean of these responses is linearly transformed to a range of 0 (worst) to 100 (best). Change from baseline is calculated as the time point value - baseline value and a decrease from baseline indicates decline in quality of life. A positive number indicates improvement in QOL.
Time Frame: Baseline and completion of chemoradiation, approximately 6-8 weeks from randomization
Population: Eligible patients enrolled after the protocol amendment who have QLQ-C30 Global Health Status score at baseline and completion of chemoradiation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 34 | 32
score on a scale | -10.3 (23.7) | -12.2 (23.5)

12. Secondary Outcome: Change From Baseline in QLQ-C30 Global Health Status Score at Completion of Post-operative Chemotherapy
Description: as for outcome 11
Time Frame: Baseline and completion of post-operative chemotherapy approximately 32 to 40 weeks from randomization based on 18 weeks of post-operative chemotherapy
Population: Eligible patients enrolled after the protocol amendment who have QLQ-C30 Global Health Status score at baseline and completion of post-operative chemotherapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 20 | 28
score on a scale | -12.5 (26.7) | -7.1 (15.0)

13. Secondary Outcome: Change From Baseline in QLQ-C30 Global Health Status Score at Two Years
Description: Global Health Status is calculated from two questions on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ]-C30. The question responses range from 1 "very poor" to 7 "excellent" such that a higher response indicates better quality of life (QOL). The mean of these responses is linearly transformed to a range of 0 (worst) to 100 (best). Change from baseline is calculated as the time point value - baseline value and a decrease from baseline indicates decline in quality of life. A negative number indicates improvement in symptoms.
Time Frame: Baseline and two years
Population: Eligible patients enrolled after the protocol amendment who have QLQ-C30 Global Health Status score at baseline and two years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 21 | 20
score on a scale | -6.8 (28.3) | -1.3 (14.4)

14. Secondary Outcome: Change From Baseline in EORTC QLQ-CR38 Gastro-intestinal Symptom Score at Completion of Chemoradiation
Description: The gastro-intestinal (GI) symptom score is calculated from five symptom questions on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ]-CR38. The question responses range from 1 (not at all) to 4 (very much) such that a higher response indicates worse symptoms. The mean of these responses is linearly transformed to a range of 0 (best) to 100 (worst). Change from baseline is calculated as the time point value - baseline value and a decrease from baseline indicates improvement in symptoms. A negative number indicates improvement in symptoms.
Time Frame: Baseline and completion of chemoradiation approximately 6-8 weeks from randomization
Population: Eligible patients enrolled after the protocol amendment who have QLQ-C38 GI score at baseline and completion of chemoradiation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 34 | 33
score on a scale | 5.9 (22.3) | 20.3 (22.1)

15. Secondary Outcome: Change From Baseline in EORTC QLQ-CR38 Gastro-intestinal Symptom Score at Completion of Post-operative Chemotherapy
Description: as for outcome 14
Time Frame: as for outcome 12
Population: Eligible patients enrolled after the protocol amendment who have QLQ-C38 GI score at baseline and completion of post-operative chemotherapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 22 | 27
score on a scale | -1.5 (12.7) | 3.9 (15.4)

16. Secondary Outcome: Change From Baseline in EORTC QLQ-CR38 Gastro-intestinal Symptom Score at Two Years
Description: as for outcome 14
Time Frame: Baseline and two years
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 21 | 20
score on a scale | 0.4 (20.3) | 6.7 (12.7)

17. Secondary Outcome: Change From Baseline in EORTC QLQ-CR38 Defecation Symptom Score at Completion of Chemoradiation
Description: The defecation symptom score is calculated from seven symptom questions on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ]-CR38. The question responses range from 1 "not at all" to 4 "very much" such that a higher response indicates worse symptoms. The mean of these responses is linearly transformed to a range of 0 (best) to 100 (worst). Change from baseline is calculated as the time point value - baseline value and a decrease from baseline indicates improvement in symptoms. A negative number indicates improvement in symptoms.
Time Frame: Baseline and completion of chemoradiation, approximately 6-8 weeks from randomization
Population: Eligible patients enrolled after the protocol amendment who have QLQ-C38 defecation score at baseline and completion of chemoradiation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 32 | 32
score on a scale | 4.8 (21.6) | 8.8 (21.8)

18. Secondary Outcome: Change From Baseline in EORTC QLQ-CR38 Defecation Symptom Score at Post-operative Chemotherapy
Description: as for outcome 17
Time Frame: Baseline and completion of post-operative chemotherapy, approximately 32 to 40 weeks from randomization based on 18 weeks of post-operative chemotherapy
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 12 | 14
score on a scale | -1.6 (16.2) | 14.6 (16.6)

19. Secondary Outcome: Change From Baseline in EORTC QLQ-CR38 Defecation Symptom Score at Two Years
Description: as for outcome 17
Time Frame: Baseline and two years
Population: Eligible patients enrolled after the protocol amendment who have QLQ-C38 defecation score at baseline and two years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Number analyzed (Participants) | 13 | 15
score on a scale | 0.4 (20.5) | -1.6 (12.9)

ADVERSE EVENTS:
Description: All eligible patients are included. Patients experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Neoadjuvant Chemoradiation With Irinotecan | Neoadjuvant Chemoradiation With Oxaliplatin
Serious Adverse Events (participants affected / at risk) | 37/70 | 36/68
Other Adverse Events (participants affected / at risk) | 70/70 | 67/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Chemoradiation With Irinotecan (N=70) | Neoadjuvant Chemoradiation With Oxaliplatin (N=68)
Blood/bone marrow - Other: (Blood and lymphatic system disorders) | 1 | 1
Hemoglobin (Blood and lymphatic system disorders) | 7 | 7
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Abdominal distention (Gastrointestinal disorders) | 0 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 3 | 3
Colitis NOS (Gastrointestinal disorders) | 0 | 2
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea NOS (Gastrointestinal disorders) | 13 | 16
Dry mouth (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Gastrointestinal - Other: (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 1
Intestinal fistula (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 5
Proctalgia (Gastrointestinal disorders) | 2 | 3
Proctitis NOS (Gastrointestinal disorders) | 0 | 3
Rectal fistula (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 2
Rectal stenosis (Gastrointestinal disorders) | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Small intestinal stricture NOS (Gastrointestinal disorders) | 3 | 4
Tooth development disorder (Gastrointestinal disorders) | 0 | 1
Vomiting NOS (Gastrointestinal disorders) | 3 | 6
Chest pain (General disorders) | 1 | 0
Death NOS (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 6
Multi-organ failure (General disorders) | 1 | 0
Pain - Other: (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 3
Rigors (General disorders) | 1 | 1
Sudden death (General disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 1
Ano-rectal infection NOS (Infections and infestations) | 0 | 1
Infection - Other: (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Blood (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Lung (pneumonia) (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Skin (cellulitis) (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Urinary tract NOS (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Wound (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Blood (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Pelvis NOS (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 1 | 0
Infection with unknown ANC: Bladder (urinary) (Infections and infestations) | 0 | 1
Peritoneal infection (Infections and infestations) | 0 | 2
Wound infection (Infections and infestations) | 0 | 1
Culture wound negative (Injury, poisoning and procedural complications) | 0 | 1
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 0 | 3
Leak (including anastomotic), GI: Small bowel (Injury, poisoning and procedural complications) | 0 | 1
Radiation recall syndrome (Injury, poisoning and procedural complications) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 3
Coagulopathy (Investigations) | 0 | 1
Leukopenia NOS (Investigations) | 8 | 5
Lymphopenia (Investigations) | 0 | 1
Metabolic/laboratory - Other: (Investigations) | 0 | 1
Neutrophil count (Investigations) | 3 | 1
Platelet count decreased (Investigations) | 2 | 3
Weight decreased (Investigations) | 1 | 3
Alkalosis NOS (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 11 | 7
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Arthritis NOS (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal/soft tissue - Other: (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3
Syncope vasovagal (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Renal failure NOS (Renal and urinary disorders) | 0 | 2
Renal/genitourinary - Other: (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Vesical fistula (Renal and urinary disorders) | 0 | 2
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Pelvic pain NOS (Reproductive system and breast disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Sweating increased (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension NOS (Vascular disorders) | 2 | 2
Thrombosis (Vascular disorders) | 2 | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Chemoradiation With Irinotecan (N=70) | Neoadjuvant Chemoradiation With Oxaliplatin (N=68)
Blood/bone marrow - Other: (Blood and lymphatic system disorders) | 1 | 5
Hemoglobin (Blood and lymphatic system disorders) | 50 | 44
Abdominal pain NOS (Gastrointestinal disorders) | 21 | 17
Constipation (Gastrointestinal disorders) | 25 | 20
Diarrhoea NOS (Gastrointestinal disorders) | 56 | 57
Dyspepsia (Gastrointestinal disorders) | 8 | 3
Faecal incontinence (Gastrointestinal disorders) | 4 | 6
Flatulence (Gastrointestinal disorders) | 8 | 4
Gastrointestinal - Other: (Gastrointestinal disorders) | 3 | 7
Hemorrhoids (Gastrointestinal disorders) | 6 | 3
Nausea (Gastrointestinal disorders) | 39 | 45
Proctalgia (Gastrointestinal disorders) | 18 | 22
Proctitis NOS (Gastrointestinal disorders) | 12 | 12
Radiation mucositis (Gastrointestinal disorders) | 3 | 4
Rectal hemorrhage (Gastrointestinal disorders) | 12 | 6
Stomatitis (Gastrointestinal disorders) | 9 | 7
Vomiting NOS (Gastrointestinal disorders) | 19 | 20
Constitutional Symptoms - Other: (General disorders) | 4 | 1
Edema: limb: (General disorders) | 3 | 7
Fatigue (General disorders) | 48 | 51
Pain - Other: (General disorders) | 5 | 5
Pyrexia (General disorders) | 4 | 6
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 17 | 14
Radiation recall syndrome (Injury, poisoning and procedural complications) | 4 | 8
Alanine aminotransferase increased (Investigations) | 18 | 27
Aspartate aminotransferase increased (Investigations) | 17 | 25
Blood alkaline phosphatase increased (Investigations) | 11 | 21
Blood bilirubin increased (Investigations) | 6 | 4
Blood creatinine increased (Investigations) | 9 | 8
Leukopenia NOS (Investigations) | 48 | 41
Lymphopenia (Investigations) | 6 | 6
Metabolic/laboratory - Other: (Investigations) | 7 | 13
Neutrophil count (Investigations) | 33 | 31
Platelet count decreased (Investigations) | 28 | 29
Weight decreased (Investigations) | 16 | 19
Anorexia (Metabolism and nutrition disorders) | 23 | 21
Dehydration (Metabolism and nutrition disorders) | 8 | 17
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 37 | 25
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 16 | 23
Hypocalcemia (Metabolism and nutrition disorders) | 15 | 22
Hypoglycemia NOS (Metabolism and nutrition disorders) | 4 | 2
Hypokalemia (Metabolism and nutrition disorders) | 18 | 24
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 7
Hyponatremia (Metabolism and nutrition disorders) | 18 | 25
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Dizziness (Nervous system disorders) | 8 | 1
Dysgeusia (Nervous system disorders) | 5 | 10
Headache (Nervous system disorders) | 2 | 4
Neuralgia NOS (Nervous system disorders) | 0 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 36 | 44
Anxiety (Psychiatric disorders) | 4 | 5
Depression (Psychiatric disorders) | 7 | 7
Insomnia (Psychiatric disorders) | 5 | 9
Bladder pain (Renal and urinary disorders) | 6 | 4
Pollakiuria (Renal and urinary disorders) | 14 | 11
Renal/genitourinary - Other: (Renal and urinary disorders) | 5 | 5
Urinary incontinence (Renal and urinary disorders) | 5 | 3
Urinary retention (Renal and urinary disorders) | 6 | 4
Erectile dysfunction NOS (Reproductive system and breast disorders) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 3
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 6 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 6
Localised exfoliation (Skin and subcutaneous tissue disorders) | 3 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4
Hypertension NOS (Vascular disorders) | 2 | 4
Hypotension NOS (Vascular disorders) | 5 | 2
Thrombosis (Vascular disorders) | 1 | 5

LIMITATIONS AND CAVEATS:
Due to excessive GI adverse events in the first 35 patients, chemotherapy dosage was modified and the protocol was amended (treatment descriptions reflect the revision). Therefore the first 35 patients are not included in outcome measure results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No